CLINICAL TRIAL: NCT04460846
Title: Evaluation of Hydration Status When Consuming Alkaline Water Compared to Reverse Osmosis Purified Water: A Randomized Controlled Cross-over Pilot Study
Brief Title: Evaluation of Hydration Status When Consuming Alkaline Water Compared to Reverse Osmosis Purified Water.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NIS165-003
Record Dates: First submitted 2020-03-11; First posted 2020-07-08 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-06

CONDITIONS: Hydration

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, cross-over trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alkaline water (Active Comparator): Participants will consume 1.5 liters per day
  Interventions: Dietary Supplement: Alkaline water
- Reverse osmosis water (Placebo Comparator): Participants will consume 1.5 liters per day
  Interventions: Dietary Supplement: Reverse osmosis water

INTERVENTIONS:
Dietary Supplement: Alkaline water — 1.5 liters per day
  Arms: Alkaline water
Dietary Supplement: Reverse osmosis water — 1.5 liters per day
  Arms: Reverse osmosis water

SUMMARY:
To conduct a randomized, double-blinded, placebo-controlled, cross-over trial in a population of chronically, moderately dehydrated people comparing two waters on hydration status.

DETAILED DESCRIPTION:
A randomized, double-blinded, placebo-controlled cross-over study design will be used to evaluate the effects of consumption of alkaline water against reverse osmosis water. The study is of 5 weeks' duration, with evaluation at baseline, 2 weeks (beginning of wash-out period), 3 weeks (end of wash-out period), and 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult people of either gender;
* Age 18 - 65 years (inclusive);
* BMI between 18.0 and 34.9 (inclusive);
* Screening results showing at least one of the following:

  * Hematocrit: Women: 45.0 or higher; Men: 48.7 or higher;
  * BUN/Creatinine ratio 20 or higher;
  * Sodium levels 146 mmol/L or higher;
  * Potassium levels 5.3 mmol/L or higher;
  * Chloride levels 108 mmol/L or higher.
* Willing to maintain a consistent diet (including medications, vitamins and supplements) and lifestyle routine throughout the study;
* Willing to abstain from coffee, tea, soft drinks, and nicotine for at least one hour prior to a clinic visit;
* Willing to abstain from alcohol for at least 12 hours prior to a clinic visit;
* Willing to maintain a consistent habit of abstaining from exercising and nutritional supplements on the morning of a study visit.

Exclusion Criteria:

* Cancer during past 12 months;
* Chemotherapy during past 12 months;
* Significant active uncontrolled illness (such as lymphoma, liver disease, kidney failure, heart failure).
* Previous major surgery to stomach or intestines [(absorption of test product may be altered) minor surgery is not a problem, including appendix and gallbladder removal];
* Implanted electronic device such as pacemaker or implantable cardioverter-defibrillator (ICD);
* Currently experiencing peripheral edema in legs and /or feet;
* Diagnosed with any blood clotting disorder or taking clotting factor concentrates;
* Diagnosis of Peripheral Artery Disease;
* Diagnosis of varicose veins;
* Currently taking blood pressure medication;
* Currently taking blood thinning medication (81mg aspirin allowed);
* Currently taking diuretic medication;
* Currently taking nutritional supplements and other substances judged by the study coordinator to negate or camouflage the effects of the test product;
* Women who are pregnant, nursing, or trying to become pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-12-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of hydration status using Bioelectrical Impedance Analysis | Change from baseline to 2 weeks
  Bioelectrical Impedance Analysis performed using an RJL system, capturing information on intracellular and extracellular water.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Jensen, PhD, Principal Investigator — NIS Labs
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States